CLINICAL TRIAL: NCT04800601
Title: Awakening of the Control of the Ankle Dorsiflexors in the Post Stroke Hemiplegic Subject to Improve Walking Activity and Social Participation: Experimental Interventional Study
Brief Title: Walking Ankle isoKinetic Exercise
Acronym: WAKE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 87RI20_0010 (WAKE)
Record Dates: First submitted 2021-03-08; First posted 2021-03-16 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Stroke Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Other: Rehabilitation program 1
- Control group (Active Comparator)
  Interventions: Other: Rehabilitation program 2

INTERVENTIONS:
Other: Rehabilitation program 1 — Both groups will benefit from a conventional rehabilitation treatment including a repetitive walking.
  In addition to this conventional rehabilitation, the experimental group will receive an ankle isokinetic program, 5 times a week, for 6 weeks (with a minimum of 25 sessions)
  Arms: Experimental group
Other: Rehabilitation program 2 — Both groups will benefit from a conventional rehabilitation treatment including a repetitive walking.
  The control group will have a supplement in conventional rehabilitation equal to the additional time of the experimental group.
  Arms: Control group

SUMMARY:
This study is a multi-center, interventional, experimental, prospective, controlled and randomized study. We propose a reeducation protocol based on an early over-solicitation of the ankle dorsiflexor muscles to promote their "awakening", limit the loss of strength associated with the functional loss and thus allow to reach a more effective walking activity. This should encourage social participation following discharge from the hospital. The main objective is to evaluate the impact of this 6 weeks program on walking speed.

DETAILED DESCRIPTION:
According to HAS, stroke is the leading cause of disability acquired in France. If 90% of patients recover walking, it is often limited with a steady speed around 0.7m/s. This limitation of walking activity is partly related to a decrease in strength associated with more or less significant spasticity. In stroke, this decrease in strength is the result of central impairment. Rehabilitation therefore involves gestural repetition. Mentiplay's review (Mentiplay et al., 2015) showing the predominance of ankle muscle strength in walking activity, we propose a protocol based on repetitive mobilization of this joint during subacute phase to promote awakening control, to limit the loss of muscle strength and thus potentiate the recovery of a more efficient walking. The strength of this study would be to verify the effectiveness of such a program in a large number of patients (5 centers involved). Its originality is to measure the impact of this program on social participation.

The patients will be recruited in 5 centers during their hospitalization, in sub-acute phase. Two groups will be formed: a control group in conventional rehabilitation; an experimental group that will perform 5x/week 300 movements of plantarflexion, dorsiflexion on isokinetic dynamometer (in passive mode, with the intention of producing the greatest possible force). This protocol will take place over 6 weeks.

Follow-up visits will take place at the end of the 6th week (which corresponds to the end of the ankle rehabilitation protocol), 6 months and one year after the beginning of the protocol.

These visits will include a clinical examination, a GaitRite carpet walking test, an isokinetic evaluation of the ankle dorsiflexor muscles strength and a SIPSO self-administered questionnaire (social participation) at 6 months and one year.

ELIGIBILITY:
Inclusion Criteria:

* First stroke,
* Ischemic or hemorrhagic stroke hospitalized in MPR in sub-acute phase (15 days to 3 months)
* Persistent deficiency of foot lifts (Medical Research Council testing: MRC <5)
* Walking alone at least 10 meters with or without technical assistance
* Absence of pain in the lower limb (EVA <2)

Exclusion Criteria:

* Cognitive or phasic disorders that do not make it possible to understand the instructions: Boston Scale BDAE <2
* Gait disorder before stroke
* Fixed stiffness of the ankle (irreducible equine less than 30 °)
* Spasticity too important: Modified Ashworth (MAS) greater than or equal to 4.
* Pregnancy or desire for pregnancy, breastfeeding
* Patient under curatorship or guardianship or under the protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
Walking speed | Week 6
  10 m walking speed measured at the end of intervention

SECONDARY OUTCOMES:
Social participation | Week 26, Week 52
  Social participation will be analyzed by specific questionnaire, the Subjective Index of Physical and Social Outcome (SIPSO) at S26 (26th week) and S52 (52th week).
Walking spatio-temporal parameters | Week 0, Week 6, Week 26, Week 52
  The parameters will be measured using a treadmill at each assessment (week 0, week 6, week 26, week 52) :
  * the duration of support phase (ms),
  * the duration of oscillating phase (ms),
  * the cadence (steps/min),
  * the step variability.
Walking speed | Week 26, Week 52
  10m speed: measured at week 26 and week 52
Dorsiflexors strength | Week 26, Week 52
  Dorsiflexors strength evaluated by isokinetic dynamometer at Week 0, Week 6, Week 26 and Week 52.
Use of technical aids to walk and the number of fall | Week 52
  The use of technical aids to walk and the number of falls will be listed in Week 52.
Correlations between walking speed /dorsiflexor muscles strength | Week 0, Week 6, Week 26, Week 52
  Correlations between walking speed /dorsiflexor muscles strength at Week 0, Week 6, Week 26 and Week 52 and walking speed/social participation at Week 26 and Week 52. (The dorsiflexor muscles strength will be evaluated by isokinetic dynamometer at Week 0, Week 6, Week 26 and Week 52. The walking speed over 10m will be measured at Week 0, Week 6, Week 26 and Week52. Social participation will be measured by questionnaire (SIPSO) at Week 26 and Week 52)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe DAVIET, Principal Investigator — University Hospital, Limoges
Locations (7):
- France (7):
  - Reeducation Institute Les Embruns, Bidart
  - University Hospital, Bordeaux
  - DUBOIS Hospital, Brive-la-Gaillarde
  - University Hospital, Limoges
  - University Institute of Rehabilitation Valmante Sud, Marseille
  - Functional rehabilitation center, Noth
  - University Hospital, Poitiers

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferry B, Compagnat M, Yonneau J, Bensoussan L, Moucheboeuf G, Muller F, Laborde B, Jossart A, David R, Magne J, Marais L, Daviet JC. Awakening the control of the ankle dorsiflexors in the post-stroke hemiplegic subject to improve walking activity and social participation: the WAKE (Walking Ankle isoKinetic Exercise) randomised, controlled trial. Trials. 2022 Aug 16;23(1):661. doi: 10.1186/s13063-022-06545-w. PMID 35974379